CLINICAL TRIAL: NCT02245464
Title: The Post Marketing Surveillance Study Conducted With a Continuous Enrollment Method to Assess Serious Adverse Events, Adverse Events, Safety, Efficacy of Micardis Tablet (Telmisartan 20, 40, 80mg p.o. Once Daily Over 2 Weeks)
Brief Title: Post Marketing Surveillance (PMS) Study to Assess Safety and Efficacy of Micardis in Patients With Essential Hypertension
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 502.479
Record Dates: First submitted 2014-09-18; First posted 2014-09-19 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients with essential hypertension
  Interventions: Drug: Telmisartan

INTERVENTIONS:
Drug: Telmisartan

SUMMARY:
The objective of this PMS study was to monitor and assess the safety of Micardis tablets in patients with hypertension over a period of 6 years

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients diagnosed with essential hypertension
* Patients without prior experience with Micardis tablet

Exclusion Criteria:

* Known hypersensitivity to Micardis tablet
* Pregnancy or breastfeeding
* Biliary atresia
* Severe hepatic failure patients
* Severe renal failure patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with essential hypertension and without prior Micardis experience
Sampling Method: Non-Probability Sample
Enrollment: 13066 (Actual)
Dates: Start 2000-11; Primary Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Blood pressure reduction | Up to 6 years
Final assessment of efficacy on a 3-point scale | Up to 6 years
Assessment of efficacy based on subject's demographics on a two-point scale | Up to 6 years
Number of patients with adverse events | Up to 6 years
Incidence rate of adverse events | Up to 6 years
  based on demographic factors
Assessment of safety on a 4-point scale | Up to 6 years
  based on adverse events and changes in abnormality of clinical laboratory tests